CLINICAL TRIAL: NCT06842342
Title: The Analgesic Effect of Ultrasound-guided Sacral Erector Spinae, Pericapsular Nerve Block and Lumber Plexus Block for Pain Relief for Hip Surgery: Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Zakarea Wfa, Lecturer of Anesthesia, Surgical ICU and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 36264PR977
Record Dates: First submitted 2025-02-08; First posted 2025-02-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Sacral Erector Block Versus Pericapsular Block Versus Lumber Plexus Block
MeSH Terms: interventions — Parapsychology; Dental Occlusion; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group LPB (Active Comparator)
  Interventions: Procedure: Lumber plexus block
- Group ESB (Active Comparator)
  Interventions: Procedure: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®)
- Group PENG (Active Comparator)
  Interventions: Procedure: PENG Block

INTERVENTIONS:
Procedure: Lumber plexus block — LPB Group: All members of this group will receive ipsilateral lumber plexus after induction of general anesthesia. The LPB will be performed by using 30 ml mixture of lidocaine 2% (10 ml), bupivacaine 0.25%(10 ml) and 10-mL normal saline will be injected at that point after repeated negative aspiration.
  Arms: Group LPB
Procedure: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®) — ESB Group: All members of this group will receive ipsilateral sacral erector spinae block after induction of general anesthesia. The ESB will be performed by using 30 ml mixture of lidocaine 2% (10 ml), bupivacaine 0.25%(10 ml) and 10-mL normal saline will be injected at that point after repeated negative aspiration.
  Arms: Group ESB
Procedure: PENG Block — PENG block: All members of this group will receive PENG block in the supine position after general anesthesia, The PENG will be performed by using 40 ml mixture of, 20 mL of 0.5 bupivacaine,10 mL of 2% lidocaine, and 10 mL of normal saline.
  Arms: Group PENG

SUMMARY:
The aim of this study to evaluate the effect of The analgesic effect of Ultrasound-guided Sacral erector spinae, Pericapsular nerve block and Lumber Plexus block for pain relief after hip surgery.

The primary outcome will be the collective morphine consumption on the 1st day post-operatively.

Secondary end points Early postoperative pain scores including static pain and passive movement pain (at PACU, at 6 ,12,18 and 24 h after surgery) will be evaluated with visual analog scale (VAS) ranging from 0 to 10, where 0 means no pain and 10 means the worst pain Intraoperative consumption of fentanyl Intraoperative adverse reactions (hypotension, bradycardia, etc.) Complications related with anesthesia (local anesthetic systemic toxicity, pneumothorax, hematoma, etc.) Performance time of block (defined as the time from ultrasound scanning to the end of injection)

DETAILED DESCRIPTION:
The hip joint connects the femur and pelvis and is responsible for multidimensional motion and mechanical stability [ 1 ]. Most hip pain is caused by the joint capsule [ 2 ]. Furthermore, the joint is largely controlled by the femoral, sciatic, and obturator nerves [ 3 ]. Patients may experience incomplete analgesia with techniques such as femoral nerve (FN) block alone due to the proximal locations of these nerves. Blocking the proximal innervation of all terminal branches innervating the hip joint (femoral, sciatic, obturator, etc.) causes significant weakness in the leg [ 1 ]. With the growth of the elderly population, more patients are undergoing hip surgeries. However, although methods are improving, no gold standard has been established for anesthesia or, more specifically, for analgesia in operations with high morbidity and high mortality [4]. Hip surgeries include hip arthroplasty (HA) (partial hip replacement, total hip replacement) and proximal femur operations (proximal femoral nailing) [5]. In fact, HA is one of the most successful orthopedic procedures in terms of improving patients' functional status and quality of life [ 6 ]. Appropriate pain management for surgical patients contributes to early mobilization, shorter hospital stays, reduced costs, and increased patient satisfaction.

Therefore, minimizing postoperative pain has become increasingly important for healthcare providers in recent years [ 7 ]. For this purpose, various analgesia techniques have been used. Although opioids typically provide effective pain relief, their use is limited due to serious side effects [ 8 ]. In recent years, peripheral nerve blocks (PNBs) have been used in the management of postoperative pain following hip surgery. The 2021 procedure-specific postoperative pain management (PROSPECT) guideline for total HA recommends several perioperative interventions to alleviate postoperative pain [9].

Erector spinae plane (ESP) block and pericapsular nerve group (PENG) block are the main safe and proven blocks used in hip operations [ 10 , 11 ]. PENG block is a novel regional analgesia technique that preserves motor function while reducing pain after HA. This technique involves injecting local anesthetic (LA) into the fascial plane between the psoas muscle and the superior pubic ramus [ 11 , 12 ].

Erector spinae plane block (ESPB) was first described as an interfascial plane block performed at the upper thoracic levels to alleviate neuropathic pain [13]. Later, its use has been reported in many thoracic procedures including mastectomy, video-assisted thoracoscopy (VATS), heart surgery, at lumbar levels for abdominal surgery, prostatectomy, lumbar spine surgery, total hip arthroplasty, and proximal femur surgery [14].

Sacral ESPB has been recently described. Case reports are showing that it is useful in various types of surgery. In case presentations, it has been reported as effective in providing analgesia in the posterior branches of the sacral nerves in pilonidal sinus surgery, in the treatment of radicular pain at the L5 - S1 level, after a sex reassignment operation hypospadias surgery, and its use in combination with lumbar ESPB for analgesia was reported after hip prosthesis surgery [15-20].

As a frequently used regional anesthesia technique for low limb surgery, lumbar plexus block (LPB) can provide effective analgesia and reduce opioid consumption for the patients undergoing total hip arthroplasty (THA) [20-22]. The lumbar plexus occasionally originates from T12 to L4. The three main branches of lumbar plexus that innervate the hip region, including the femoral, obturator, and lateral femoral cutaneous nerve, can be blocked with a single-level LPB at L3 [21] observed the spread of local anesthetic with MRI in the volunteers underwent LPB at L4. The injectate was mainly confined between L2 and L4 and barely diffused to T12-L1. Thus, insufficient of analgesia of the incision area may occur due to the failure block of the branches derive from T12 and L1, such as iliohypogastric and subcostal nerve [23]. As we know, the effect of regional block depends on the coverage of related nerve branches at the surgical area. Therefore, to provide a more comprehensive coverage on the wide range of lumbar plexus, multiple-level block techniques, e.g., LPB at L2 and L3, at L3 and L4, or even combined with T12 L1 paravertebral block (PVB), were applied in some studies [24-27]. However, it is conceivable that these expert techniques may require more operator expertise, consume more performance time, increase the discomfort of the patients, and have a greater risk of complications [ 28-32]. Thus, a both effective and convenient method should be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years old without cognitive dysfunction

  * Body mass index (BMI) between 18.5 and 30 kg/m 2 and the weight ≥ 50 kg
  * American Society of Anesthesiologists (ASA) classification I-II

Exclusion Criteria:

* Refuse to general anesthesia (GA) with tracheal intubation

  * Nerve block is contraindicated due to various reasons, such as open trauma, hematoma or skin infection at the blocking area, lower limb neuro-muscular disorders
  * Coagulation dysfunction or anticoagulation therapy
  * Known hypersensitivity or allergy to local anesthetics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Morphine consumption over 24 hours | 24 hours postoperatively
  will be the collective morphine consumption on the 1st day post-operatively

SECONDARY OUTCOMES:
Pain score | During and after operation within 24 hours
  Early postoperative pain scores including static pain and passive movement pain (at PACU, at 6 ,12,18 and 24 h after surgery) will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta, Tanta, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided